CLINICAL TRIAL: NCT02058290
Title: A Pain Relief Trial Utilizing the Infiltration of a Multivesicular Liposome Formulation of Bupivacaine, EXPAREL(R): A Phase 4 Health Economic Trial in Adult Patients Undergoing Laparoscopic Colectomy (IMPROVE-Lap Colectomy)
Brief Title: A Health Economic Trial in Adult Patients Undergoing Laparoscopic Colectomy
Acronym: IMPROVE-Lap
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slower than expected enrollment
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MA402S23B6A/6B; NCT01460485 (obsolete NCT alias); NCT01461122 (obsolete NCT alias); NCT01461135 (obsolete NCT alias); NCT01509820 (obsolete NCT alias); NCT01534988 (obsolete NCT alias); NCT01963975 (obsolete NCT alias)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Bowel Obstruction
Keywords: laparoscopic colectomy
MeSH Terms: conditions — Intestinal Obstruction | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Morphine Sulfate or Sponsor-approved Equivalent (Active Comparator): Standard of Care (SOC)
  Interventions: Drug: IV morphine sulfate or Sponsor-approved equivalent
- EXPAREL (Experimental): EXPAREL (bupivacaine liposome injectable suspension)
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: IV morphine sulfate or Sponsor-approved equivalent — Patients in this group will receive IV morphine sulfate or Sponsor-approved equivalent via a patient-controlled analgesia (PCA) pump, as needed. The PCA pump will be set up postsurgically as soon as possible and prior to the patient leaving the post-anesthesia care unit (PACU) or immediately upon transfer to a floor if the stay in the PACU is less than one hour.
  Arms: IV Morphine Sulfate or Sponsor-approved Equivalent
Drug: EXPAREL — Patients will receive 266 mg EXPAREL diluted with preservative-free 0.9% normal saline to a total volume of 40 cc administered via wound infiltration prior to wound closure. When not contraindicated, 30 mg IV ketorolac will be given at the end of surgery. If not indicated, an IV non-steroidal anti-inflammatory drug (NSAID) may be substituted per the site's standard of care.
  All patients will be offered rescue analgesia, as needed.
  Other Names: bupivacaine liposome injectable suspension
  Arms: EXPAREL

SUMMARY:
This study is designed to compare the standard of care against EXPAREL (bupivacaine liposome injectable suspension) to determine if total opioid consumption is reduced when using EXPAREL, therefore possibly reducing total hospital costs.

DETAILED DESCRIPTION:
This is a Phase 4, prospective, sequential, open-label study designed to evaluate the efficacy, safety, and health economic benefits of intraoperative local wound infiltration with EXPAREL (bupivacaine liposome injectable suspension) compared with postsurgical administration of standardized intravenous (IV) morphine sulfate or Sponsor-approved equivalent for postsurgical analgesia in adult patients undergoing laparoscopic colectomy with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age.
* Patients scheduled to undergo laparoscopic segmental colectomy with planned primary anastamosis, as defined by cecectomy, right hemicolectomy, resection of transverse colon, left hemicolectomy, or sigmoidectomy. (Note: patients who converted from a planned laparoscopic colectomy to an open colectomy were not eligible.)
* Ability to provide informed consent, adhere to study visit schedule, and complete all study assessments.

Exclusion Criteria:

* Patients with a history of hypersensitivity or idiosyncratic reactions or intolerance to any local anesthetic, opioid, or propofol.
* Patients who abuse alcohol or other drug substance.
* Patients with severe hepatic impairment.
* Patients currently pregnant or who may become pregnant during the course of the study or who are unwilling to use acceptable means of contraception for at least 1 month before and 1 month after dosing. Acceptable means of contraception include hormonal contraceptives (e.g., oral, injectable, implantable), effective barrier methods (e.g., condoms with spermicide), intrauterine device, lifestyle with a personal choice of abstinence, non-heterosexual lifestyle, or in a strictly monogamous relationship with a partner who has had a vasectomy.
* Patients with any psychiatric, psychological, or other condition that the Investigator feels may make the patient an inappropriate candidate for this clinical study.
* Participation in an EXPAREL study within the last 30 days.
* Patients who have received any investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the patient's participation in this study.

In addition, a patient was ineligible if he or she met the following criteria during surgery:

* Patients who had any concurrent surgical procedure.
* Patients with unplanned multiple segmental resections of large intestine.
* Patients who converted from laparoscopic-assisted colectomy to traditional open colectomy.
* Patients who had unplanned, temporary or permanent colostomies, ileostomies, or the like placed.
* Patients who received intraoperative administration of opioids (other than fentanyl or analogs) or any other analgesic, local anesthetics, or anti-inflammatory agents.
* Patients who received Entereg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Lee, MD, Principal Investigator — Albany Medical College; Keith Candiotti, MD, Principal Investigator — University of Miami; Sergio Bergese, MD, Principal Investigator — Ohio State University; Eric M Haas, MD, Principal Investigator — The Methodist Hospital Research Institute; Jorge Marcet, MD, Principal Investigator — Tampa General Hospital; Anjali Kumar, MD, Principal Investigator — Medstar Health Research Institute
Locations (6):
- United States (6):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami, Dept. Anesthesiology, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Albany Medical College, Albany, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Cohen SM, Vogel JD, Marcet JE, Candiotti KA. Liposome bupivacaine for improvement in economic outcomes and opioid burden in GI surgery: IMPROVE Study pooled analysis. J Pain Res. 2014 Jun 24;7:359-66. doi: 10.2147/JPR.S63764. eCollection 2014. PMID 25018650

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Morphine Sulfate or Sponsor-approved Equivalent: Standard of Care (SOC)
  IV morphine sulfate or Sponsor-approved equivalent: Patients in this group received IV morphine sulfate or Sponsor-approved equivalent via a patient-controlled analgesia (PCA) pump, as needed. The PCA pump was set up postsurgically as soon as possible and prior to the patient leaving the post-anesthesia care unit (PACU) or immediately upon transfer to a floor if the stay in the PACU was less than one hour.
- EXPAREL: EXPAREL (bupivacaine liposome injectable suspension)
  EXPAREL: Patients received 266 mg EXPAREL diluted with preservative-free 0.9% normal saline to a total volume of 40 cc administered via wound infiltration prior to wound closure. When not contraindicated, 30 mg IV ketorolac was given at the end of surgery. If not indicated, an IV non-steroidal anti-inflammatory drug (NSAID) could be substituted per the site's standard of care.
  All patients were offered rescue analgesia, as needed.
Period: Overall Study
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL
Started | 77 | 45
Completed | 66 | 36
Not Completed | 11 | 9
Not completed — Protocol Violation | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Didn't meet intraoperative criteria | 8 | 7
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 122 subjects were enrolled. Of these, 105 subjects received study drug: 67 subjects received IV morphine sulfate or sponsor-approved equivalent and 38 subjects received EXPAREL.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL | Total
Number analyzed (Participants) | 67 | 38 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.35) | 57.8 (11.86) | 58.3 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 21 | 56
  Male | 32 | 17 | 49
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 60 | 34 | 94
American Society of Anesthesiologist (ASA) Classification [Number; unit: participants]
  Normal [1] | 1 | 0 | 1
  Mild Systemic Disease [2] | 32 | 25 | 57
  Severe Systemic Disease [3] | 32 | 13 | 45
  Severe Systemic Disease Threat to Life [4] | 2 | 0 | 2
Patient's Pain Level 24 Hours Prior to Surgery [Mean (Standard Deviation); unit: units on a scale] — Patient's Pain Level 24 Hours Prior to Surgery was measured on a scale from 0 to 10 where 0 = no pain and 10 = worst possible pain.
  units on a scale | 1.9 (2.14) | 1.3 (0.86) | 1.7 (1.81)

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Burden
Description: Total opioid consumed (IV and PO) postsurgically until hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: Of the 77 subjects who were enrolled in Group 1, 56 were included in the efficacy analysis set. Of the 45 subjects who were enrolled in Group 2, 26 were included in the efficacy analysis set.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL
Number analyzed (Participants) | 56 | 26
mg | 96.47 (77.74) | 32.06 (53.16)
Statistical Analysis 1: Comparison: IV Morphine Sulfate or Sponsor-approved Equivalent vs EXPAREL; Test type: Superiority or Other; p < 0.0001, ANOVA

2. Primary Outcome: Health Economic Benefits - Total Cost of Hospitalization
Description: Total cost of hospitalization until the time hospital discharge order is written or through Day 30, whichever was sooner.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL
Number analyzed (Participants) | 56 | 26
dollars | 15158.79 (11417.50) | 14802.70 (18382.12)
Statistical Analysis 1: Comparison: IV Morphine Sulfate or Sponsor-approved Equivalent vs EXPAREL; Test type: Superiority or Other; p = 0.2612, ANOVA

3. Primary Outcome: Health Economic Benefits - Length of Stay (LOS)
Description: Length of stay, recorded in days, defined as the time of completion of the wound closure until the hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure at time hospital discharge order is written or Day 30, whichever is sooner
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL
Number analyzed (Participants) | 56 | 26
days | 4.0 [0 to 30] | 3.0 [1.9 to 10.7]
Statistical Analysis 1: Comparison: IV Morphine Sulfate or Sponsor-approved Equivalent vs EXPAREL; Test type: Superiority or Other; p = 0.0019, Log Rank

4. Secondary Outcome: Incidence of Opioid-related Adverse Events
Description: Incidence of opioid-related adverse events defined as somnolence, respiratory depression, hypoventilation, hypoxia, dry mouth, nausea, vomiting, constipation, sedation, confusion, pruritus, urinary retention, and postoperative ileus.
Time Frame: Wound closure at time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL
Number analyzed (Participants) | 56 | 26
participants | 23 | 2

5. Secondary Outcome: Patient Satisfaction With Pain Treatment After Surgery
Description: Responses to question pertaining to patient satisfaction with pain treatment
Time Frame: Wound closure at time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL
Number analyzed (Participants) | 56 | 26
participants
  Extremely Satisfied | 30 | 17
  Satisfied | 19 | 5
  Neither Satisfied nor Dissatisfied | 0 | 2
  Dissatisfied | 3 | 0
  Extremely Dissatisfied | 1 | 0
  Not Reported | 3 | 2

ADVERSE EVENTS:
Time Frame: Through Day 30 post surgery.
Description: Of the 122 subjects enrolled, the safety analysis set included 67 subjects from Group 1 and 38 subjects from Group 2.
Arm/Group | IV Morphine Sulfate or Sponsor-approved Equivalent | EXPAREL
Serious Adverse Events (participants affected / at risk) | 9/67 | 5/38
Other Adverse Events (participants affected / at risk) | 53/67 | 15/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Morphine Sulfate or Sponsor-approved Equivalent (N=67) | EXPAREL (N=38)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 1
Clostridial Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Wound Infection (Infections and infestations) | 0 | 1
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 1
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stent Placement (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Blood Urea Nitrogen (BUN) Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
White Blood Cells Increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Morphine Sulfate or Sponsor-approved Equivalent (N=67) | EXPAREL (N=38)
Anemia (Blood and lymphatic system disorders) | 4 | 2
Leukocytosis (Blood and lymphatic system disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 2 | 2
Abdominal Distention (Gastrointestinal disorders) | 5 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 23 | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Chest Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 1
Cellulitis (Infections and infestations) | 0 | 2
Clostridial Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 2 | 1
Blood Pressure Increased (Investigations) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 7 | 0
Hypoethesia (Nervous system disorders) | 2 | 0
Confusional State (Psychiatric disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 5 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No